CLINICAL TRIAL: NCT07321522
Title: Early Introduction and Sustained Ingestion (EISI) Using Two Educational Opportunities - A Pilot Study
Brief Title: Early Introduction and Sustained Ingestion (EISI) Using Two Educational Opportunities in Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, R. Sharon Chinthrajah, Professor of Medicine, Pulmonary Allergy and Critical Care Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 81307
Record Dates: First submitted 2025-12-15; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): The participants will be provided with three sets of educational materials to learn about early introduction of food allergens.
- Enhanced Educational Opportunities (Experimental): The participants will be provided with three sets of educational materials to learn about early introduction of food allergens, as well as 3 in-person monthly teaching sessions (up to 3 months), lasting 30 minutes to enhance the information and allow for questions. This arm will also have one to two in-clinic feedings of any of the top 9 most allergenic foods. The oral feeding portion will add an additional 1 to 2 hours at the one of the 3 visits.
  Interventions: Behavioral: Educational Sessions and Opportunities on Early Introduction and Sustained Ingestion; Behavioral: In person feeding session

INTERVENTIONS:
Behavioral: Educational Sessions and Opportunities on Early Introduction and Sustained Ingestion — The participant will attend three in person sessions on the basics of food allergy, food allergy reactions, feeding safety and readiness, fiber, ultra processed foods, diet diversity, and advancing food textures in the infant diet. The educational sessions will last 20 - 30 minutes every month for three months.
  Arms: Enhanced Educational Opportunities
Behavioral: In person feeding session — Participants will attend an in-person feeding of a known top 9 food allergen (hen's egg, cow's milk, peanut, tree nuts, soy, wheat, fin fish, shellfish, and sesame) to the infant at least one time, and up to two times. The clinic feeding will last 1 - 2 hours.
  Arms: Enhanced Educational Opportunities

SUMMARY:
The objective of the study is to see whether early feeding of potentially allergic foods can be increased with educational materials alone or with educational materials and additional in-person support opportunities. This study will help guide what types of support pediatricians and allergists give to new parents.

DETAILED DESCRIPTION:
This 6 month study will randomly assign caretaker/child dyads into two groups; 50% will be assigned to the intervention group, the other 50% to the standard-of-care group. Using the foods of each families home and culture, participants in the standard-of-care group will be instructed through 3 packets metered one month apart of scientifically supported written, audio and video materials that are widely available to the general public. The intervention group will receive the same educational materials at the same time points as the standard-of-care group. The intervention group will additionally have in-person or live-stream video opportunities instructing further about the same materials and ask questions of the research team. The intervention group will additionally have one and up to two opportunities to feed their infant in the clinical research unit one of the top 9 known US allergenic foods (Top 9) with the feeding staffed with emergency response personnel and supportive clinical care. Both groups will complete the same quiz following each educational set of materials to evaluate the helpfulness and understanding of each. Both groups will record the intake of the Top 9 for the first 3 months. Both groups will record the intake of the Top 9, fruit/vegetable, whole grains, legumes, seeds and ultra processed food intake for the second 3 months of the study. Both groups will undergo a blood draw on the infant at the first and last visits. Both groups will complete a pre and post study questionnaire.

The standard-of-care group will be offered the opportunity to return to the clinic to feed a Top 9 food when their enrollment is fully completed.

ELIGIBILITY:
Inclusion Criteria for both Infant and Caregiver/Parent Participants

* Born term (37 weeks - 41 weeks gestation)
* Infants with or without a family history of allergic disease
* Infants with or without mild to moderate eczema
* Infants who have not yet started consuming T9 foods (excluding cow's milk or soy if it is in their infant formula)
* Parent or caregiver ≥ 18 years of age
* Agree to infant blood draw (two)
* Agree to participate in the 6 month research study

Exclusion Criteria:

* Infants with a physician confirmed food allergy
* Infants who do not eat fully by an oral route such as tube-fed or tube-supplemented babies
* Infants with developmental delay
* Infants with severe eczema
* Infants who are already consuming Top 9 known allergenic foods
* Infants participating in another study looking at diet, oral immunotherapy or the use of a biological agent

Ages: 4 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Compare the infant age at which allergenic foods were introduced | Baseline up to six months.
  The average age of introduction of allergenic foods will be calculated and compared between groups.
Compare the allergenic food intake frequency. | At the start of intervention and month 1, month 2, month 3, month 4, month 5 and month 6.
  The participants will self report how many times they took a particular allergenic food each month. This outcome will be compared between the two groups.
Compare the quantity of allergenic foods consumed. | At the start of intervention and month 4, month 5 and month 6.
  The participants will measure the amount of allergenic foods consumed daily as either: a taste, ≤ 1 teaspoon,
  1 - 2 teaspoons or ≥ 3 tablespoons. The total amount of food consumed in a month will be compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Chinthrajah, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warren CM, Aktas ON, Manalo LJ, Bartell TR, Gupta RS. The epidemiology of multifood allergy in the United States: A population-based study. Ann Allergy Asthma Immunol. 2023 May;130(5):637-648.e5. doi: 10.1016/j.anai.2022.12.031. Epub 2022 Dec 31. PMID 36596337
- [Background] Gupta R, Holdford D, Bilaver L, Dyer A, Holl JL, Meltzer D. The economic impact of childhood food allergy in the United States. JAMA Pediatr. 2013 Nov;167(11):1026-31. doi: 10.1001/jamapediatrics.2013.2376. PMID 24042236
- [Background] Togias A, Cooper SF, Acebal ML, Assa'ad A, Baker JR Jr, Beck LA, Block J, Byrd-Bredbenner C, Chan ES, Eichenfield LF, Fleischer DM, Fuchs GJ 3rd, Furuta GT, Greenhawt MJ, Gupta RS, Habich M, Jones SM, Keaton K, Muraro A, Plaut M, Rosenwasser LJ, Rotrosen D, Sampson HA, Schneider LC, Sicherer SH, Sidbury R, Spergel J, Stukus DR, Venter C, Boyce JA. Addendum guidelines for the prevention of peanut allergy in the United States: Report of the National Institute of Allergy and Infectious Diseases-sponsored expert panel. J Allergy Clin Immunol. 2017 Jan;139(1):29-44. doi: 10.1016/j.jaci.2016.10.010. PMID 28065278
- [Background] Du Toit G, Roberts G, Sayre PH, Bahnson HT, Radulovic S, Santos AF, Brough HA, Phippard D, Basting M, Feeney M, Turcanu V, Sever ML, Gomez Lorenzo M, Plaut M, Lack G; LEAP Study Team. Randomized trial of peanut consumption in infants at risk for peanut allergy. N Engl J Med. 2015 Feb 26;372(9):803-13. doi: 10.1056/NEJMoa1414850. Epub 2015 Feb 23. PMID 25705822
- [Background] Perkin MR, Logan K, Marrs T, Radulovic S, Craven J, Flohr C, Lack G; EAT Study Team. Enquiring About Tolerance (EAT) study: Feasibility of an early allergenic food introduction regimen. J Allergy Clin Immunol. 2016 May;137(5):1477-1486.e8. doi: 10.1016/j.jaci.2015.12.1322. Epub 2016 Feb 17. PMID 26896232
- [Background] Natsume O, Kabashima S, Nakazato J, Yamamoto-Hanada K, Narita M, Kondo M, Saito M, Kishino A, Takimoto T, Inoue E, Tang J, Kido H, Wong GW, Matsumoto K, Saito H, Ohya Y; PETIT Study Team. Two-step egg introduction for prevention of egg allergy in high-risk infants with eczema (PETIT): a randomised, double-blind, placebo-controlled trial. Lancet. 2017 Jan 21;389(10066):276-286. doi: 10.1016/S0140-6736(16)31418-0. Epub 2016 Dec 9. PMID 27939035
- [Background] Venter C, Groetch M. Emerging concepts in introducing foods for food allergy prevention. Curr Opin Clin Nutr Metab Care. 2025 May 1;28(3):263-273. doi: 10.1097/MCO.0000000000001126. Epub 2025 Mar 7. PMID 40072493
- [Background] Berni Canani R, Carucci L, Coppola S, D'Auria E, O'Mahony L, Roth-Walter F, Vassilopolou E, Agostoni C, Agache I, Akdis C, De Giovanni Di Santa Severina F, Faketea G, Greenhawt M, Hoffman K, Hufnagel K, Meyer R, Milani GP, Nowak-Wegrzyn A, Nwaru B, Padua I, Paparo L, Diego P, Reese I, Roduit C, Smith PK, Santos A, Untersmayr E, Vlieg-Boerstra B, Venter C. Ultra-processed foods, allergy outcomes and underlying mechanisms in children: An EAACI task force report. Pediatr Allergy Immunol. 2024 Sep;35(9):e14231. doi: 10.1111/pai.14231. PMID 39254357
- [Background] Boden S, Lindam A, Venter C, Ulfsdotter RL, Domellof M, West CE. Diversity of complementary diet and early food allergy risk. Pediatr Allergy Immunol. 2025 Jan;36(1):e70035. doi: 10.1111/pai.70035. PMID 39868464
- [Background] Harbottle Z, Malm Nilsson E, Venter C, Golding MA, Ekstrom S, Protudjer JLP. Parental Motivation for Introducing Babies' First Foods and Common Food Allergens. Nutrients. 2025 May 27;17(11):1812. doi: 10.3390/nu17111812. PMID 40507081
- [Background] Samady W, Warren C, Bilaver LA, Zaslavsky J, Jiang J, Gupta R. Early Peanut Introduction Awareness, Beliefs, and Practices Among Parents and Caregivers. Pediatrics. 2023 Aug 1;152(2):e2022059376. doi: 10.1542/peds.2022-059376. PMID 37476922
- [Background] Smith HG, Nimmagadda S, Gupta RS, Warren CM. Food allergen introduction practices and parent/caregiver attitudes based on family history of food allergy. Front Allergy. 2025 Mar 19;6:1562667. doi: 10.3389/falgy.2025.1562667. eCollection 2025. PMID 40176928
- See also: The Health Belief Model of Behavior Change — http://www.ncbi.nlm.nih.gov/books/NBK606120/